CLINICAL TRIAL: NCT06799936
Title: A Communication-Priming Intervention to Improve Shared Decision-Making Between Older Adults With Advanced Chronic Kidney Disease and Clinicians: A Cluster-Randomized Controlled Trial
Brief Title: A Communication-Priming Intervention to Improve Shared Decision-Making Between Older Adults With Advanced CKD and Clinicians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, YUEN Jacqueline Kwan Yuk, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17609724
Record Dates: First submitted 2025-01-27; First posted 2025-01-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5
Keywords: Communication; Priming; Decision-making; Older adults; Chronic kidney disease; CKD-Priming Jumpstart
MeSH Terms: conditions — Renal Insufficiency, Chronic; Communication

STUDY DESIGN:
Intervention Model Description: The Study Model includes two components for priming intervention, for patients and clinicians respectively:
  Patients: Patients will complete a "CKD Jumpstart- Tips" communication priming tool before a target clinic visit. Within one week prior to and on the day of the visit, patients will receive a "CKD Jumpstart- Tips" patient summary sheet.
  Clinicians: Within one week prior to and on the day of the target clinic visit, clinicians will receive a "CKD Jumpstart- Tips" clinician priming sheet which contains an abstracted version of the patients' survey responses and communication tips tailored to the patient's responses.
  Patients in the control group will receive usual care (e.g. education classes and information on kidney failure treatment options). Clinicians in the control group will provide consultations to patients under usual practices.
  Clinicians will be randomized at a 1:1 ratio to the intervention or control group with stratification by study site.
Who Masked: Outcomes Assessor
Masking Description: The statistical analyst will be blinded to site and arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Priming Intervention arm (Experimental): Patients in the priming intervention arm will be provided and are expected to complete the "CKD Jumpstart- Tips" communication priming tool prior to a target clinic visit.
  Within one week prior to and on the day of the target clinic visit, patients will receive a "CKD Jumpstart- Tips" patient summary sheet which includes a summary of survey responses that can be shared with their healthcare team and tips on communication with clinician during upcoming visit.
  Clinicians in the priming intervention arm will receive a "CKD Jumpstart- Tips" clinician priming sheet in the patient's medical chart within one week prior to and on the day of the target clinic visit. The priming sheet includes an abstracted version of the patients' survey responses and communication tips tailored to the patient's responses based on Vitaltalk curricular materials.
  Interventions: Other: "CKD Jumpstart- Tips" priming intervention
- Usual care arm (No Intervention): Additional education classes and information in written or multimedia formats reviewing kidney failure treatment options will be made available per routine care and will not be dictated by the study. Patients will be asked whether they have attended an education session or provided informational materials at baseline.

INTERVENTIONS:
Other: "CKD Jumpstart- Tips" priming intervention — The intervention includes 2 components:
  1. Patient Priming: Patients will receive the "Jumpstart CKD- Tips" communication priming tool within 1 week before and on the day of a target clinic visit, which includes surveys on (i) Understanding of illness and possible treatment options, (ii) Readiness for treatment discussion and information preferences, (iii) Health priorities, goals, and preferences (iv) Preferred roles in decision-making. The "Jumpstart CKD- Tips" patient priming sheet includes (a) A summary of their survey responses that can be shared with their healthcare team, and (b) Tips on communication with clinician during upcoming visit.
  2. Clinician Priming: Within 1 week before and on the day of the target clinic visit, clinicians will receive a "Jumpstart CKD- Tips" clinician priming sheet which contains (a) An abstracted version of the patients' survey responses and (b) Communication tips tailored to the patient's responses based on Vitaltalk curricula materials.
  Arms: Priming Intervention arm

SUMMARY:
To achieve the goal of reaching consensus about the preferred treatment option that best aligns with the goals and values of patients, the investigators developed a 'CKD Jumpstart- Tips" priming tool tailored for older adults with advanced CKD that is based on communication principles from VitalTalk and Elwyn's goal-based SDM model.

The investigators hypothesize that compared with patients in the usual care group, patients in the 'CKD Jumpstart- Tips' intervention group will have:

1. increased level of shared decision-making (observer-based and patient-reported),
2. improved quality of communication,
3. increased patient involvement in decision-making,
4. lower decisional conflict,
5. lower decision regret,
6. decreased time to decision,
7. improved adherence to treatment choice, and
8. improved health-related quality-of-life.

DETAILED DESCRIPTION:
To enhance the communication on shared decision-making between older adults with advanced kidney disease and clinicians, the investigator's research team developed the "CKD Jumpstart- Tips" communication-priming intervention.

This study aims to conduct a cluster-randomized controlled trial to assess the effects of the 'CKD Jumpstart- Tips' communication-priming intervention on shared decision-making between older adults with advanced kidney disease and their clinicians.

The primary objective of the study is to evaluate the effects of the intervention on observer-based shared decision-making in the target consultation.

The secondary objective is to evaluate the effects of intervention on patient-reported shared decision-making, quality of communication, patient involvement in decision-making, decisional conflict, decision regret, timing of and adherence to treatment choice, and health-related quality of life. Consultation length will also be captured as a process measure.

ELIGIBILITY:
Inclusion criteria for the two groups of participants (i.e. Clinicians and Patients):

1. Clinicians

   - Nephrology specialists or higher physician trainees who provide specialty care to older adults with advanced chronic kidney disease
2. Patients

   * Diagnosis of advanced CKD Stage 4 or 5 (eGRF <30 ml/min)
   * Chinese- or English-speaking
   * Identified as patient with whom their clinician plans to discuss advanced kidney disease treatment options in the upcoming clinic visit
   * Able to provide written informed consent and complete questionnaires
   * Can be contacted by phone

Exclusion criteria for patients:

* Patients will be excluded if they are eligible for kidney transplant, currently on dialysis, or lack decision-making capacity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Observer-rated shared decision making | T1 (Immediately after target visit)
  Observer-rated shared decision making will be measured using the validated 5-item OPTION5 instrument based on Collaborative Deliberation. Each item is scored on a 0 (no effort) to 4 (exemplary effort) scale. Two raters will complete an online training module from the OPTION5 developers and then undergo calibration training through assessing five audio-recordings of consultations with other trained study team members. The two raters will independently rate audio-recordings of the target visit, and then compare ratings and resolve discrepancies by consensus. The final item scores will be added for a summary score ranging from 0 to 20 and a scale score ranging from 0 to 100. Higher total scores imply higher degrees of SDM.

SECONDARY OUTCOMES:
Patient-reported shared decision-making | T1 (Immediately after target visit)
  Patient-reported shared decision-making will be measured using the Chinese-validated 9-item SDM-Q-9 after the target visit. Patients will rate the items on a scale from 0 (Completely disagree) to 5 (Completely Agree). Total scores range from 0 to 100. The higher the score, the higher the perception of SDM. The SDM-Q-9 showed a high reliability with a high internal consistency (Cronbach's α > 0.9) and item discrimination.
Quality of Communication | T1 (Immediately after target visit)
  Quality of Communication will be assessed using the Chinese version of the patient-reported Quality of Communication questionnaire (QOC-C). The QOC-C was previously validated by the investigator's team in advanced CKD patients to assess patients' perception of the quality of clinician communication on end-of-life care issues and has a 3-factor structure. The investigators will administer the illness trajectory (4 items) and end-of-life care planning subscales (6 items) and the two summary items. Each item rates the clinician's skill on a scale from 0 ("very worst I can imagine") to 10 ("very best I can imagine").
Consultation time | T1 (Immediately after target visit)
  Consultation time will be assessed from audio-recordings of the target clinic visit consultations.
Patient involvement in decision-making | T1 (Immediately after target visit)
  Patient involvement in decision-making will be measured using the 1-item validated modified Control Preferences Scale (CPS). The CPS consists of 1 item with five response options, each corresponding to a description of the patient's role in decision-making. The score representing these role descriptions ranges from 1 to 5, from 1 indicating the patient making the treatment decisions, 3 indicating the patient making the decisions jointly with the physician, to 5 indicating the physician making the decisions. The CPS has shown good reliability and validity.
Decisional conflict | T1 (Immediately after target visit), T2 (3 Months), T3 (6 Months)
  Decisional conflict will be measured using the Chinese validated 16-item Decisional Conflict scale (DCS). The DCS covers five subscales measuring how well informed patients feel about their choices and associated benefits and risks, clarity of values, support received in decision making, level of uncertainty about the best choice, and perceived effectiveness of decision making. Each item is rated on a five-point Likert scale. The total score is calculated by averaging the sum of the items and then multiplying by 25. The total score ranges from 0 to 100, with a higher score indicating more decisional conflict. The Chinese version has good internal consistency, with Cronbach's α of 0.81.
Decisional regret | T2 (3 Months), T3 (6 Months)
  Decisional regret will be measured using the Chinese validated five-item Decision Regret scale (DRS). The DRS measures distress or remorse after a health care decision. Each item is rated on a five-point Likert scale. The total score is calculated by averaging the sum of the five items and then multiplying by 25. The total score ranges from 0 to 100, with a higher score indicating greater decision regret. The Chinese version has good internal consistency with Cronbach's α of 0.83.
Timing of and adherence to treatment choice | T1 (Immediately after target visit), T2 (3 Months), T3 (6 Months)
  Timing of and adherence to treatment choice will be assessed by patient report and by chart review. Patients will be asked whether and when they have indicated their treatment choice and any changes in their treatment choice. Chart abstraction from the medical record will occur at the end of data collection period to assess for clinician documentation of the initial treatment choice and any subsequent change in treatment choice. The timing and setting of the documentation will also be recorded.
Health-related quality of life | T2 (3 Months), T3 (6 Months)
  Health-related quality of life will be assessed using the validated Chinese version of the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal). The FACIT Pal is a patient-reported measure of health-related quality of life (QOL) for patients with advanced illness. It contains four domains: physical (7 items), social/family (7 items), emotional (6 items) and functional (7) wellbeing and a Palliative care subscale (PalS, 19 items). Each item is rated from 0 (not at all) to 4 (very much). Higher scores reflect higher QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline KY Yuen, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared in order to protect patient privacy. However, summary data of patients will be shared upon reasonable request to the study's Principal Investigator"

REFERENCES:
- [Background] Zhou X, Tian X, Fan Y, Sun M, Wang Z, Huang Y, Xiao W. Psychometric Properties of the Chinese Version of the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal) in Patients With Advanced Cancer. J Pain Symptom Manage. 2024 Jan;67(1):e8-e15. doi: 10.1016/j.jpainsymman.2023.09.020. Epub 2023 Sep 26. PMID 37769823
- [Background] Xu RH, Zhou LM, Wong EL, Wang D, Chang JH. Psychometric Evaluation of the Chinese Version of the Decision Regret Scale. Front Psychol. 2020 Dec 3;11:583574. doi: 10.3389/fpsyg.2020.583574. eCollection 2020. PMID 33424697
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Lam WW, Kwok M, Liao Q, Chan M, Or A, Kwong A, Suen D, Fielding R. Psychometric assessment of the Chinese version of the decisional conflict scale in Chinese women making decision for breast cancer surgery. Health Expect. 2015 Apr;18(2):210-20. doi: 10.1111/hex.12021. Epub 2012 Nov 21. PMID 23167846
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Elwyn G, Vermunt NPCA. Goal-Based Shared Decision-Making: Developing an Integrated Model. J Patient Exp. 2020 Oct;7(5):688-696. doi: 10.1177/2374373519878604. Epub 2019 Oct 17. PMID 33294602
- [Background] McCaffery KJ, Holmes-Rovner M, Smith SK, Rovner D, Nutbeam D, Clayman ML, Kelly-Blake K, Wolf MS, Sheridan SL. Addressing health literacy in patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S10. doi: 10.1186/1472-6947-13-S2-S10. Epub 2013 Nov 29. PMID 24624970
- [Background] Sepucha KR, Borkhoff CM, Lally J, Levin CA, Matlock DD, Ng CJ, Ropka ME, Stacey D, Joseph-Williams N, Wills CE, Thomson R. Establishing the effectiveness of patient decision aids: key constructs and measurement instruments. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S12. doi: 10.1186/1472-6947-13-S2-S12. Epub 2013 Nov 29. PMID 24625035
- [Background] Davis JL, Davison SN. Hard choices, better outcomes: a review of shared decision-making and patient decision aids around dialysis initiation and conservative kidney management. Curr Opin Nephrol Hypertens. 2017 May;26(3):205-213. doi: 10.1097/MNH.0000000000000321. PMID 28212179
- [Background] Morton R. Do Dialysis Decision Aids Improve Treatment Decision-Making? Perit Dial Int. 2016 Jul-Aug;36(4):359-61. doi: 10.3747/pdi.2016.00017. No abstract available. PMID 27385805
- [Background] Jungers P, Zingraff J, Albouze G, Chauveau P, Page B, Hannedouche T, Man NK. Late referral to maintenance dialysis: detrimental consequences. Nephrol Dial Transplant. 1993;8(10):1089-93. PMID 8272221
- [Background] Hughes SA, Mendelssohn JG, Tobe SW, McFarlane PA, Mendelssohn DC. Factors associated with suboptimal initiation of dialysis despite early nephrologist referral. Nephrol Dial Transplant. 2013 Feb;28(2):392-7. doi: 10.1093/ndt/gfs431. Epub 2012 Dec 4. PMID 23222418
- [Background] Davison SN. End-of-life care preferences and needs: perceptions of patients with chronic kidney disease. Clin J Am Soc Nephrol. 2010 Feb;5(2):195-204. doi: 10.2215/CJN.05960809. Epub 2010 Jan 14. PMID 20089488
- [Background] Berkhout-Byrne N, Gaasbeek A, Mallat MJK, Rabelink TJ, Mooijaart SP, Dekker FW, van Buren M. Regret about the decision to start dialysis: a cross-sectional Dutch national survey. Neth J Med. 2017 Jul;75(6):225-234. PMID 28741581
- [Background] Ladin K, Lin N, Hahn E, Zhang G, Koch-Weser S, Weiner DE. Engagement in decision-making and patient satisfaction: a qualitative study of older patients' perceptions of dialysis initiation and modality decisions. Nephrol Dial Transplant. 2017 Aug 1;32(8):1394-1401. doi: 10.1093/ndt/gfw307. PMID 27576590
- [Background] Song MK, Lin FC, Gilet CA, Arnold RM, Bridgman JC, Ward SE. Patient perspectives on informed decision-making surrounding dialysis initiation. Nephrol Dial Transplant. 2013 Nov;28(11):2815-23. doi: 10.1093/ndt/gft238. Epub 2013 Jul 30. PMID 23901048
- [Background] Hussain JA, Flemming K, Murtagh FE, Johnson MJ. Patient and health care professional decision-making to commence and withdraw from renal dialysis: a systematic review of qualitative research. Clin J Am Soc Nephrol. 2015 Jul 7;10(7):1201-15. doi: 10.2215/CJN.11091114. Epub 2015 May 5. PMID 25943310
- [Background] Morton RL, Tong A, Howard K, Snelling P, Webster AC. The views of patients and carers in treatment decision making for chronic kidney disease: systematic review and thematic synthesis of qualitative studies. BMJ. 2010 Jan 19;340:c112. doi: 10.1136/bmj.c112. PMID 20085970
- [Background] Verberne WR, Konijn WS, Prantl K, Dijkers J, Roskam MT, van Delden JJM, Bos WJW. Older patients' experiences with a shared decision-making process on choosing dialysis or conservative care for advanced chronic kidney disease: a survey study. BMC Nephrol. 2019 Jul 16;20(1):264. doi: 10.1186/s12882-019-1423-x. PMID 31311511
- [Background] Frazier R, Levine S, Porteny T, Tighiouart H, Wong JB, Isakova T, Koch-Weser S, Gordon EJ, Weiner DE, Ladin K. Shared Decision Making Among Older Adults With Advanced CKD. Am J Kidney Dis. 2022 Nov;80(5):599-609. doi: 10.1053/j.ajkd.2022.02.017. Epub 2022 Mar 26. PMID 35351579
- [Background] Waldron T, Carr T, McMullen L, Westhorp G, Duncan V, Neufeld SM, Bandura LA, Groot G. Development of a program theory for shared decision-making: a realist synthesis. BMC Health Serv Res. 2020 Jan 23;20(1):59. doi: 10.1186/s12913-019-4649-1. PMID 31973754
- [Background] Stiggelbout AM, Pieterse AH, De Haes JC. Shared decision making: Concepts, evidence, and practice. Patient Educ Couns. 2015 Oct;98(10):1172-9. doi: 10.1016/j.pec.2015.06.022. Epub 2015 Jul 15. PMID 26215573
- [Background] Galla JH. Clinical practice guideline on shared decision-making in the appropriate initiation of and withdrawal from dialysis. The Renal Physicians Association and the American Society of Nephrology. J Am Soc Nephrol. 2000 Jul;11(7):1340-1342. doi: 10.1681/ASN.V1171340. No abstract available. PMID 10864592
- [Background] Cheung AK, Chang TI, Cushman WC, Furth SL, Hou FF, Ix JH, Knoll GA, Muntner P, Pecoits-Filho R, Sarnak MJ, Tobe SW, Tomson CRV, Lytvyn L, Craig JC, Tunnicliffe DJ, Howell M, Tonelli M, Cheung M, Earley A, Mann JFE. Executive summary of the KDIGO 2021 Clinical Practice Guideline for the Management of Blood Pressure in Chronic Kidney Disease. Kidney Int. 2021 Mar;99(3):559-569. doi: 10.1016/j.kint.2020.10.026. PMID 33637203
- [Background] Jassal SV, Watson D. Dialysis in late life: benefit or burden. Clin J Am Soc Nephrol. 2009 Dec;4(12):2008-12. doi: 10.2215/CJN.04610709. Epub 2009 Nov 5. PMID 19965545
- [Background] Tang SC. CKD prevention: Perspectives in Hong Kong. Nephrology (Carlton). 2018 Oct;23 Suppl 4:72-75. doi: 10.1111/nep.13468. PMID 30298664
- [Background] Xie Y, Bowe B, Mokdad AH, Xian H, Yan Y, Li T, Maddukuri G, Tsai CY, Floyd T, Al-Aly Z. Analysis of the Global Burden of Disease study highlights the global, regional, and national trends of chronic kidney disease epidemiology from 1990 to 2016. Kidney Int. 2018 Sep;94(3):567-581. doi: 10.1016/j.kint.2018.04.011. Epub 2018 Aug 3. PMID 30078514
- See also: The communication tips used in the "CKD Jumpstart- Tips" intervention were based on VitalTalk curricular materials. — https://www.vitaltalk.org/